CLINICAL TRIAL: NCT04097457
Title: A Community-implemented, Parent-mediated, Group Intervention for Children With Autism Spectrum Disorder (ASD) and Disruptive Behaviors.
Brief Title: Group Based Parent Training for Children With Autism and Disruptive Behaviors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Eyal Cohen, Study coordinator, Hebrew University of Jerusalem
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GroupPT ASD
Record Dates: First submitted 2019-09-16; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Butter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parent mediated intervention (PMI) group (Experimental): A short term parent training protocol based on behavioral principles, which is delivered by trained therapists. The protocol includes eleven core sessions, a home visit session, follow-up telephone booster sessions and seven supplemental sessions, designed to be delivered to parents in an outpatient and home settings. The protocol is administered to groups of 4 families.
  Interventions: Behavioral: "Parent training for disruptive behaviors" manual (Bearss, Johnson, Handen, Butter, Lecavalier, Smith & Scahill, 2018)
- Waitlist control (Experimental): Families will be recruited and will fill out measure for 3 months prior to participation and will then join the active intervention
  Interventions: Behavioral: "Parent training for disruptive behaviors" manual (Bearss, Johnson, Handen, Butter, Lecavalier, Smith & Scahill, 2018)
- Individual (Experimental): A short term parent training protocol based on behavioral principles, which is delivered by trained therapists. The protocol includes eleven core sessions, a home visit session, follow-up telephone booster sessions and seven supplemental sessions, designed to be delivered to parents in an outpatient and home settings. In this arm the protocol is administered individually to families.
  Interventions: Behavioral: "Parent training for disruptive behaviors" manual (Bearss, Johnson, Handen, Butter, Lecavalier, Smith & Scahill, 2018)

INTERVENTIONS:
Behavioral: "Parent training for disruptive behaviors" manual (Bearss, Johnson, Handen, Butter, Lecavalier, Smith & Scahill, 2018) — The intervention is a short term parent training program based on behavioral principles, which can be delivered by trained therapist. The manual includes eleven core sessions, home visit session, follow-up telephone booster sessions and seven supplemental sessions, designed to be delivered individually to parents in an outpatient setting.
  The protocol will be administered to groups of 3-4 parents, with a quantitative pretest-post test design evaluated at five time points, including a follow up at one month post intervention. The protocol will be administered in various community and educational locations, such as schools and community centers

SUMMARY:
The goal of the study is to providing parents of children diagnosed with autism spectrum disorders (ASD) and disruptive behaviors essential skills to manage their children's behaviors using an evidence based parent training protocol. Beyond the feasibility of delivering an evidence based intervention in groups and with community partners, primary and secondary outcomes in both the children and the parents who participated in the study are assessed during and after the intervention process

DETAILED DESCRIPTION:
the investigators will deliver parent-mediated, community-implemented, group intervention for parents of young children with autism and disruptive behavior. The intervention is 11-12 weeks and will take place in community settings such as special education schools and community centers.

Within these meetings parents will be given the skills to understand their child's behavior and work to modify those that are clinically disruptive to the child and their environment.

Groups will be facilitated by student therapists under direct weekly supervision of a Board Certified Behavior Analyst (BCBA). Data will be collected before, after, and throughout the intervention, primarily by parent-report with one teacher-report measure and two (pre/post) filmed parent-child interactions.

The primary desired outcome is a measurable decrease in the child's disruptive behaviors and an increase in their adaptive behaviors. Although the intervention specifically targets disruptive behavior, we expect to see consequent improvement in a number of linked domains. These represent desired secondary outcomes.

First, as a result of receiving concrete skills and seeing improvement in their child's behavior, as well as due to participation in the group with other families, a reduction in parental stress and an increase in their perceived self-efficacy should occur, as well as a reduction in the stress of the non-participating parent.

Second, after the reduction in disruptive behaviors there should be an improvement in autism symptomatology. Improvements in behavior will allow the child to benefit more from their environments, leading to social and developmental gains.

In the context of the current study, the impact of the intervention on family accommodation is also assessed, hypothesizing that by learning how to analyse and modify behaviors, parents are gaining a broader insight into the impact their own behaviors have on that of their children.

ELIGIBILITY:
Inclusion Criteria:

* Formal ASD diagnosis

Exclusion Criteria:

-

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-09-02 (Estimated); Study Completion 2021-01-02 (Estimated)

PRIMARY OUTCOMES:
The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects (Aman, M. G., Singh, N. N., Stewart, A. W., & Field, C. J.,1985) | Administered to parents and teachers at baseline, 4 weeks, 8 weeks, 12 weeks (end-point), 16 weeks and 20 weeks (follow-up). The measure will be administered at different time points to follow changes in severe disruptive behaviors of the participants
  A caregiver and teacher report measure of disruptive behaviors including 58 items, each rated on a four-point Likert scale (0-3), with higher scores indicative of more severe problem behavior. Includes five subscales: Irritability (tantrums, aggression and self-injury, 15 items); Social Withdrawal (16 items); Stereotypic Behavior (7 items); Hyperactivity (16 items); and Inappropriate Speech (4 items). In children with ASD, the ABC subscales demonstrate adequate internal consistencies (α=.77-.94) and convergent validity (Kaat, Lecavalier, & Aman, 2014).
  The measure will be administered at different time points on order to follow changes in the disruptive behaviors of the participants.
Home Situations Questionnaire (HSQ) (Barkley & Murphy, 1998) | Administered to parents at baseline, 12 weeks and at 20 weeks.The measure will be administered at different time points in order to follow changes in compliance levels of the participants.
  A caregiver-rated scale for child noncompliance across 24 everyday situations. Each item is rated as a problem: ''yes'' or ''no''; ''yes'' items are then scored from 1 (mild) to 9 (severe), on two subscales: 'Demand-Specific' and 'Socially Inflexible' (Chowdhury et al. 2010). The total severity score is divided by 24 to obtain a per item mean.
Social Responsiveness Scale (SRS) (Constantino & Gruber, 2005) | Administered to parents at baseline, 12 weeks and at 20 weeks. The measure will be administered at different time points in order to follow changes in social-related behaviors of the participants.
  A caregiver - and teacher-report measure of child social competence with 65 items, each rated on a four-point Likert scale (1-4), with higher scores indicative of more problematic social-related behaviors, in the domains of social awareness, social cognition, social communication, social motivation, and autistic mannerisms (e.g., restricted or repetitive behaviors). All subscales have acceptable internal consistency (α = .77-.92) and test-retest reliability (Constantino et al., 2003)
Adaptive Behavior Assessment System (ABAS-II) | administered to participating parents at baseline, 12 weeks and at 20 weeks. The measure will be administered at different time points in order to follow changes related to adaptive behaviors of the participants.
  A comprehensive evaluation tool, covering the ten adaptive behavior deficit areas defined by the DSM-5 (APA, 2013), and it is recommended for use as part of the standard ASD diagnostic evaluation process, by the Ministry of Health in Israel. The ABAS-II provides standard scores on the following core domains: Communication; Use of Community Resources; Academic Functional Skills; Daily Living Skills; Health and Security; Leisure; Self-Help; Self-Direction; Socialization and Occupation, as well as a General Adaptive Behavior Composite Score (GAC). Items are rated on a four-point Likert scale (0-3), with higher scores indicative of higher adaptive functioning.

SECONDARY OUTCOMES:
Parenting Stress Index Short Version (PSI-SR) (Abidin, 1990) | administered to all participating and non-participating parents at baseline, 12 weeks and at 20 weeks.The measure will be administered at different time points in order to follow changes in stress levels of parent participants.
  A self-report inventory designed to measure the overall level of parenting stress an individual is experiencing and it examine stressors associated specifically with the parental role and do not include stresses associated with other life roles and events. The PSI-SR has strong psychometric properties and has been used in a number of studies of autism and parent training, and was also found valid and reliable when tested on Israeli parents (sharf 1989; Turkel 2002). It contains 36 items, each rated on a five-point Likert scale (1-5), with higher scores indicative of more parenting stress and includes Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI) and Difficult Child (DC) sub-scales.

CONTACTS AND LOCATIONS:
Overall Officials: Judah Koller, PsyD, Principal Investigator — Hebrew University in Jerusalem
Locations (1):
- The Hebrew university, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bearss K, Johnson C, Handen B, Smith T, Scahill L. A pilot study of parent training in young children with autism spectrum disorders and disruptive behavior. J Autism Dev Disord. 2013 Apr;43(4):829-40. doi: 10.1007/s10803-012-1624-7. PMID 22941342
- [Background] Bearss K, Johnson C, Smith T, Lecavalier L, Swiezy N, Aman M, McAdam DB, Butter E, Stillitano C, Minshawi N, Sukhodolsky DG, Mruzek DW, Turner K, Neal T, Hallett V, Mulick JA, Green B, Handen B, Deng Y, Dziura J, Scahill L. Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: a randomized clinical trial. JAMA. 2015 Apr 21;313(15):1524-33. doi: 10.1001/jama.2015.3150. PMID 25898050
- [Background] Bearss K, Lecavalier L, Minshawi N, Johnson C, Smith T, Handen B, Sukhodolsky D, Aman M, Swiezy N, Butter E, Scahill L. Toward an exportable parent training program for disruptive behaviors in autism spectrum disorders. Neuropsychiatry (London). 2013 Apr;3(2):169-180. doi: 10.2217/npy.13.14. PMID 23772233
- [Background] Michelson D, Davenport C, Dretzke J, Barlow J, Day C. Do evidence-based interventions work when tested in the "real world?" A systematic review and meta-analysis of parent management training for the treatment of child disruptive behavior. Clin Child Fam Psychol Rev. 2013 Mar;16(1):18-34. doi: 10.1007/s10567-013-0128-0. PMID 23420407
- See also: Protocol — https://www.rubinetwork.org/